CLINICAL TRIAL: NCT05139888
Title: A Pilot Study Evaluating the Feasibility and Usability of ToeFX Light Therapy Device for Mild to Moderate Distal Subungual Onychomycosis (DSO) of the Toenail
Brief Title: Light Therapy for Onychomycosis Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ToeFX Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TFX-LTS-001
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Onychomycosis of Toenail

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to two different groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single wavelength light (red) only (Experimental): Arm 1 will test the core technology of the ToeFX system; this study reproduces methods well-described in the literature. After application of the formulation, nails affected by onychomycosis are exposed to red light at a wavelength of 630-660 nm intensity of 200 mW/cm2.
  Interventions: Device: Single wavelength light (red) only
- Dual wavelength light (red/blue) (Experimental): Some research has shown that exposure to mild blue light can have anti-inflammatory effects that would improve patient onychomycosis outcomes. We will assess whether inclusion of blue light in the protocol affects the clinical outcome.
  Interventions: Device: Dual wavelength light (red/blue)

INTERVENTIONS:
Device: Single wavelength light (red) only — Clinicians should confirm a diagnosis of distal subungual onychomycosis (DSO). Clinician should assign an OSI score to each nail using the Onychomycosis Severity Index (OSI). The ToeFX system is intended for use in any room in which standard foot care treatments are routinely administered. Debridement should not be carried out more proximally than the most proximal margin of the dystrophic nail, as this can interfere with assessment of clear nail area attributable to the device intervention. The clinician should debride the nail, apply formula, and position the affected foot directly under the ToeFX ClearToe Therapy red light (640-660 nm). For safety, the light has a built-in timer and automatically switches off after 15 minutes. The process should be repeated every 2 weeks for 6 months.
  Arms: Single wavelength light (red) only
Device: Dual wavelength light (red/blue) — Clinicians should confirm a diagnosis of distal subungual onychomycosis (DSO). Clinician should assign an OSI score to each nail using the Onychomycosis Severity Index (OSI). The ToeFX system is intended for use in any room in which standard foot care treatments are routinely administered. Debridement should not be carried out more proximally than the most proximal margin of the dystrophic nail, as this can interfere with assessment of clear nail area attributable to the device intervention. The clinician should debride the nail, apply formula, and position the affected foot directly under the ToeFX ClearToe Therapy dual wavelength light (640-660 nm and 405-450 nm). For safety, the light has a built-in timer and automatically switches off after 15 minutes. The process should be repeated every 2 weeks for 6 months..
  Arms: Dual wavelength light (red/blue)

SUMMARY:
This is a pilot prospective study designed to capture information about the safety and effectiveness of the ToeFX Therapy Light.

DETAILED DESCRIPTION:
According to a report published by the NCBI on January 14, 2015, some 3 to 12% of the population is affected by toenfail fungus, with older populations more likely to be affected. Indeed, fungal infection of nails (onychomycosis) is among the most prevalent infectious diseases in humans. According to a communication released by the Ontario College of Physicians and Surgeons in September 2019, the cure rate for topical treatments is only 6-23% after 1 year. Even after 1 year of treatment, topical treatments have limited efficacy. Moreover, onychomycosis is cosmetically distressing.

This study will be an open-label, prospective pilot study. The subjects will be 100 patients who suffer from distal subungual onychomycosis. The purpose of the study is to establish the efficacy of the ToeFX Therapy Light, which has shown compelling results in in vitro and ex vivo (cadaver) studies but has not been tested in patients. Specifically, the investigators wish to:

1. Determine the safety and efficacy of this therapy in the treatment of distal subungual onychomycosis of the toenail.
2. Determine the number of treatments required to clear the nail and to cure the fungus.
3. Finalize the treatment protocol, device design and user interface.
4. Test re-infection or recurrence of fungus post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* have a clinical diagnosis of mild to moderate DSO in the nail of at least one great toe, with 20% to 50% clinical involvement of the target toenail, without dermatophytomas or lunula (matrix) involvement, without lunular or proximal involvement.
* exhibit positive mycology results (i.e., KOH test and culture of a dermatophyte) from the target great toenail, confirming common dermatophytes such as T. rubrum.
* are willing to refrain from using polish or other medication on treated toenails or on the skin immediately adjacent to the toenails during the treatment period unless directed to do so by the investigator.
* are willing to refrain from using topical steroids or topical antifungals on toenails or the skin immediately adjacent to the toenails or systemic antifungals for the duration of the study.
* are willing to provide signed and dated written voluntary informed consent in English before any protocol-specific procedures are performed.
* are able to complete the study and comply with study instructions.

Exclusion Criteria:

* females who are pregnant, plan to become pregnant during the study, or are nursing a child.
* persons who are hypersensitive to topical creams, ointments, medications, or surfactants.
* persons who have received systemic antifungal therapy for any reason within 3 months, or topical antifungal therapy on the toenails or skin immediately adjacent to the toenails within 3 weeks prior to the start of the study.
* persons who have received an investigational drug within 4 weeks of the first dose of study product, or who are scheduled to receive an investigational drug other than the study product during the study.
* persons who have participated in a clinical trial for the systemic treatment of onychomycosis of the toenails within 6 months prior to the first dose of study product.
* persons who are not prepared to give up use of any nail cosmetic products for the duration of the study.
* persons who have any known immunodeficiency or history of malignancy in the last 4 years, excluding nonmelanoma skin cancer.
* persons currently suffering from any disease or condition, that could include abnormal laboratory tests, and/or who are currently using medication which in the opinion of the investigator may affect the evaluation of the study product or place the subject at undue risk.
* persons with psoriasis, lichen planus, or other medical conditions known to induce nail changes, other abnormalities or can causes of nail breakdown that can predispose to secondary fungal infection. Trauma from ill-fitting shoes, running, or overly aggressive nail care can also induce changes visually indistinguishable from onychomycosis that could result in a clinically abnormal toenail.
* patients with glucose-6 phosphate dehydrogenase (G6PD) deficiency or hypersensitivity/allergies to methylene blue
* persons with a history of any condition that could possibly affect absorption of drug (e.g., gastrectomy), uncontrolled diabetes, clinically significant peripheral vascular disease or peripheral circulatory impairment, or has had any major illness within 30 days prior to the screening examination.
* persons with a history of drug, prescription medicine, or alcohol abuse within the past 2 years.
* smokers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2024-12-19 (Estimated); Study Completion 2024-12-19 (Estimated)

PRIMARY OUTCOMES:
An increase in healthy new nail growth free of fungal infection ("clear nail"), 6-12 months post-treatment | 1 year
  The investigators will monitor whether participants attain
  * at least 6 mm increase in clear nail, or
  * an additional 60 mm2 of clear nail, or
  * complete clearance 6 months after the first treatment if less than 6 mm distal nail was involved prior to treatment.
  The investigators will verify by taking a photograph prior to every treatment to assess the change in millimeters (mm) of clear nail. Millimeters of clear nail from the base of the toenail will be determined from digital photographs. An increase in "clear nail" between the two points indicates that the toenail has improved and is positive for study success. A decrease in mm of clear nail between the two points indicates that the toenail has worsened and is negative for study success. Length of the unaffected part of the target nail is measured in mm along the midpoint from the nail fold to the proximal border of the affected part (lowest point affected) along the midpoint of the nail.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rabinovich, MD, Principal Investigator — McMaster University
Locations (1):
- Hewak Foot Clinic, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No